CLINICAL TRIAL: NCT01670045
Title: A Multi-national, Multi-center Non-interventional Study in Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab
Brief Title: A Non-Interventional Study of RoActemra/Actemra (Tocilizumab) in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28216
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Results first posted 2016-05-10 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rheumatoid Arthritis Participants: Participants with moderate to severe rheumatoid arthritis (RA) according to the American College of Rheumatology (ACR) criteria and the Disease Activity Score based on 28 Joint Count (DAS28) who were on tocilizumab treatment within 8 weeks prior to start of study will receive tocilizumab in accordance with the licensed label recommendations, and will be observed for 6 months. The study is designed as non-interventional, no additional intervention in terms of follow-up visit, complementary examination or medication is required.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab in accordance with the licensed label recommendation.

SUMMARY:
This multi-center observational study will evaluate the use and efficacy of RoActemra/Actemra (tocilizumab) in patients with moderate to severe rheumatoid arthritis. Eligible patients initiated on RoActemra/Actemra treatment according to the licensed label will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis according to the revised (1987) ACR criteria
* Patient in whom the treating physician has made the decision to commence RoActemra/Actemra treatment in accordance with the local label (DMARD-IR, TNF-IR or need of RoActemra/Actemra monotherapy); this can include patients who have received RoActemra/Actemra treatment within 8 weeks prior to the enrolment visit

Exclusion Criteria:

* Patients who have received RoActemra/Actemra more than 8 weeks prior to the enrolment visit
* Patients who have previously received RoActemra/Actemra in a clinical trial or for compassionate use
* Patients who have received treatment with an investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* Patients with a history of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis initiating treatment with RoActemra/Actemra
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Indonesia (9):
  - Balikpapan
  - Bandung
  - Central Jakarta
  - Central Java
  - Denpasar
  - Jakarta
  - Malang
  - Manado
  - Medan

RESULTS

PARTICIPANT FLOW:
Groups:
- Rheumatoid Arthritis Participants: Participants with moderate to severe rheumatoid arthritis (RA) according to the American College of Rheumatology (ACR) criteria and the Disease Activity Score Based on 28 Joint Count (DAS28) who were on tocilizumab treatment within 8 weeks prior to start of study received tocilizumab in accordance with the licensed label recommendations, were observed for 6 months. The study was designed as non-interventional, no additional intervention in terms of follow-up visit, complementary examination or medication was required.
Period: Overall Study
Arm/Group | Rheumatoid Arthritis Participants
Started | 43
Completed | 27
Not Completed | 16
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 11

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants who received at least one dose of tocilizumab.
Groups:
- Rheumatoid Arthritis Participants: Participants with moderate to severe RA according to the ACR criteria and the DAS28 who were on tocilizumab treatment within 8 weeks prior to start of study received tocilizumab in accordance with the licensed label recommendations, were observed for 6 months. The study was designed as non-interventional, no additional intervention in terms of follow-up visit, complementary examination or medication was required.
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
Age, Continuous [Mean (Full Range); unit: years] | 44 [18 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Remained on Tocilizumab Treatment at 6 Months After Treatment Initiation
Time Frame: Month 6
Population: ITT.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
percentage of participants | 63

2. Secondary Outcome: Percentage of Participants With RA Diagnosis
Description: Percentage of participants was reported based on the timing RA was diagnosed. Timings included more than 5 years, less than 5 years. Participants with unknown timing were reported under "unknown".
Time Frame: Baseline up to Day 5
Population: ITT.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
percentage of participants
  More than 5 years | 39.5
  Less than 5 years | 55.8
  Unknown | 4.6

3. Secondary Outcome: Percentage of Participants With Different Body Mass Index (BMI)
Description: BMI was calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2). BMI from 16 to 18.5 = underweight, BMI from 18.5 to 25= normal weight, BMI from 25 to 30= overweight, BMI from 30 to 40 = obese.
Time Frame: Baseline up to Day 5
Population: ITT.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
percentage of participants
  Underweight | 25.6
  Normal weight | 39.5
  Overweight | 14
  Obese | 20.9

4. Secondary Outcome: Percentage of Participants With Rheumatoid Factor Status
Description: Percentage of participants with rheumatoid factor status was reported as "positive" or "negative".
Time Frame: Baseline up to Day 5
Population: ITT.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
percentage of participants
  Positive | 41.9
  Negative | 58.1

5. Secondary Outcome: Percentage of Participants With Anti-Citrullinated Cyclic Peptide (Anti-CCP) Status
Description: Percentage of participants with anti-CCP status were reported as "positive", negative" and "unknown".
Time Frame: Baseline up to Day 5
Population: ITT.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
percentage of participants
  Positive | 81.4
  Negative | 11.6
  Unknown | 7

6. Secondary Outcome: Percentage of Participants With a Reduction of at Least 2.6 Units in DAS28 From Baseline
Description: The DAS28 score is a measure of the participants' disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], participant's global assessment (PtGA) of disease activity [visual analog scale (VAS): 0 millimeter (mm)=no disease activity to 100 mm=maximum disease activity] and the erythrocyte sedimentation rate (ESR). DAS28 was calculated using following formulas: DAS28-ESR = 0.56*square root (sqrt) (TJC28) + 0.28*sqrt(SJC28) + 0.70*natural logarithm (ln) (ESR) + 0.014*PtGA of disease activity. A total possible score of 0 to approximately 10, with higher score indicating worse disease activity. A reduction of at least 2.6 units from Baseline in DAS28 was considered as significant clinical improvement.
Time Frame: Baseline, Month 1, 2, 3, 4, 5, 6
Population: ITT.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
percentage of participants
  Month 1 | 6.8
  Month 2 | 12.5
  Month 3 | 25.6
  Month 4 | 41.7
  Month 5 | 55.9
  Month 6 | 63

7. Secondary Outcome: Number of Participants Achieving a Response According to European League Against Rheumatism (EULAR) Criteria
Description: Response was determined using EULAR criteria based upon DAS28 absolute scores at the assessment visit and the DAS28 improvement from Baseline. Participants with a score less than or equal to (≤) 3.2 and DAS28 improvement of greater than (>) 1.2 points were assessed as having a 'good' response. Participants with a score ≤3.2 and DAS28 improvement of >0.6 to ≤1.2 points, score of >3.2 and ≤5.1 with DAS28 improvement of >0.6 to ≤1.2 points, score of >3.2 and ≤5.1 with DAS28 improvement of >1.2 points, score of >5.1 and DAS28 improvement of >1.2 points were assessed as having a 'moderate' response. Participants with a score ≤3.2 and DAS28 improvement of ≤ 0.6 points, score of >3.2 and ≤5.1 with DAS28 improvement of ≤ 0.6 points, score of >5.1 and DAS28 improvement of >0.6 to ≤1.2 points, score of >5.1 and DAS28 improvement of ≤ 0.6 points were assessed as having a 'no' response.
Time Frame: Baseline up to Month 6
Population: ITT.
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
participants
  Good response | 23
  Moderate response | 16
  No response | 4

8. Secondary Outcome: Number of Participants With Different Types of Simplified Disease Activity Index (SDAI)
Description: The SDAI was calculated as [SJC (28 joints) + TJC (28 joints) + VAS patient global assessment of disease activity + VAS physician global assessment of disease activity+CRP level(milligram/deciliter {mg/dL})]. VAS assessments: 0 centimeters (cm)=no disease activity to 10 cm=maximum disease activity'. Scores ranged from 0 to 86, with higher scores also indicating increased disease activity. SDAI score ≤ 3.3 is 'remission', score > 3.3 and ≤ 11 is 'low disease activity', score > 11 and ≤ 26 is 'moderate disease activity', score > 26 is 'high disease activity'. SDAI was reported as 'not available' for participants with no data on physical/patient global assessment of disease activity.
Time Frame: Baseline up to Month 6
Population: ITT.
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
participants
  Remission | 1
  Low disease activity | 19
  Moderate disease activity | 10
  High disease activity | 4
  Not available | 9

9. Secondary Outcome: Number of Participants With Different Types of Clinical Disease Activity Index (CDAI)
Description: The CDAI was calculated as [SJC (28 joints) + TJC (28 joints) + VAS patient global assessment of disease activity + VAS physician global assessment of disease activity]. VAS assessments: 0 cm =no disease activity to 100 cm=maximum disease activity'. CDAI scores ranged from 0 to 76, with higher scores indicating increased disease activity. CDAI score ≤ 2.8 is 'remission', score > 2.8 and ≤ 10 is 'low disease activity', score > 10 and ≤ 22 is 'moderate disease activity', score > 22 is 'high disease activity'. CDAI was reported as 'not available' for participants with no data on physical/patient global assessment of disease activity.
Time Frame: Baseline up to Month 6
Population: ITT.
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
participants
  Remission | 1
  Low disease activity | 19
  Moderate disease activity | 11
  High disease activity | 3
  Not available | 9

10. Secondary Outcome: Percentage of Participants Achieving a Response According to ACR Criteria
Description: ACR20/50/70 percent (%) response is defined as a ≥ 20%/50%/70% improvement (reduction) compared with baseline for both TJC28 and SJC28, as well as for three of the additional five ACR core set variables: Participant's assessment of pain over the previous 24 hours: using a VAS, left end of the line 0 cm=no pain to right end of the line 10 cm=unbearable pain; Patient's global assessment of disease activity and physician's global assessment of disease activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; health assessment questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or erythrocyte sedimentation rate].
Time Frame: Month 1, 2, 3, 4, 5, 6
Population: ITT.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
percentage of participants
  ACR20: Month 1 | 16.7
  ACR20: Month 2 | 48.7
  ACR20: Month 3 | 65.8
  ACR20: Month 4 | 75.0
  ACR20: Month 5 | 84.8
  ACR20: Month 6 | 84.6
  ACR50: Month 1 | 4.8
  ACR50: Month 2 | 15.4
  ACR50: Month 3 | 31.6
  ACR50: Month 4 | 61.2
  ACR50: Month 5 | 63.7
  ACR50: Month 6 | 65.3
  ACR70: Month 1 | 2.4
  ACR70: Month 2 | 0.0
  ACR70: Month 3 | 7.9
  ACR70: Month 4 | 30.6
  ACR70: Month 5 | 48.5
  ACR70: Month 6 | 53.8

11. Secondary Outcome: Number of Participants With Reduction/Withdrawal of Disease-modifying Anti-rheumatic Drugs (DMARDs) and/or Corticosteroids
Description: Participants with reduction/withdrawal of DMARDs and corticosteroids at baseline (before trial period) and up to Month 6 (during trial period) were reported.
Time Frame: Baseline, up to Month 6
Population: ITT.
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
participants
  DMARDS: Baseline | 16
  DMARDS: up to Month 6 | 1
  Corticosteroid: Baseline | 1
  Corticosteroid: up to Month 6 | 1

12. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity at Months 3 and 6
Description: Physician's global assessment of disease activity over the previous 24 hours was assessed using a VAS where left end of the line 0 mm=no disease activity to right end of the line 100 mm=maximum disease activity.
Time Frame: Baseline, Months 3, 6
Population: ITT. Here "number of participants analyzed" included evaluable participants for the outcome measure and "n" included evaluable participants at specified time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 36
mm
  Month 3 (n=36) | -29 (3.11)
  Month 6 (n=0) | NA (NA) — Data was not reported as there were no evaluable participants for this time point.

13. Secondary Outcome: Percentage of Participants With Tocilizumab Dose Modifications
Time Frame: Baseline up to Month 6
Population: ITT.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 43
percentage of participants | 33

ADVERSE EVENTS:
Time Frame: Baseline up to Month 6
Groups:
- Rheumatoid Arthritis Participants: Participants with moderate to severe RA and the DAS28 joint scores who were on tocilizumab treatment within 8 weeks prior to start of study received tocilizumab in accordance with the licensed label recommendations, were observed for 6 months. The study was designed as non-interventional, no additional intervention in terms of follow-up visit, complementary examination or medication was required.
Arm/Group | Rheumatoid Arthritis Participants
Serious Adverse Events (participants affected / at risk) | 14/43
Other Adverse Events (participants affected / at risk) | 3/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis Participants (N=43)
Diarrhea (Gastrointestinal disorders) | 2
Febris (General disorders) | 1
Severe pain (General disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Gastropathy (Gastrointestinal disorders) | 2
Dry Gangrene (General disorders) | 1
Left below knee lower limb amputation (General disorders) | 1
Popliteal artery thrombosis (Vascular disorders) | 1
Severe breakthrough back pain (General disorders) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis Participants (N=43)
Neutropenia (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.